CLINICAL TRIAL: NCT02156661
Title: Oxytocin and Emotion Processing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXT-FC-14
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Healthy Males
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator): Oxytocin: Syntocinon-Spray, Novartis
  intranasal administration, 24 IU oxytocin; ; 3 puffs per nostril, each with 4 IU OXT
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin

SUMMARY:
The purpose of this study is to determine whether oxytocin influences emotional processing and learning of emotional and social stimuli.

DETAILED DESCRIPTION:
An effect of OXT on emotion processing and anxiety has been broadly investigated in animal studies. However, in humans, effects seem more complex.

The rationale of the study is to examine direct effects of OXT to processing and learning of emotional and social values in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Current or past psychiatric disease
* Current or past physical illness
* Psychoactive medication
* Tobacco smokers
* MRI contraindication

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Brain activity | During emotion processing
  fMRI

SECONDARY OUTCOMES:
Psychophysiological response | During stimuli presentation
  Skin conductance response